CLINICAL TRIAL: NCT02994420
Title: Steroid Hormones in the Peripheral and Central Control of Eating in Women - Physiological Reactions to Eating in Normal- and Overweight Women
Brief Title: Endocrine and Neural Control of Eating in Women
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-0525
Record Dates: First submitted 2016-08-11; First posted 2016-12-15 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Normal Body Weight; Obesity
Keywords: Obesity; Menstrual Cycle; Gonadal Steroid Hormones; Satiety Response; Glucagon-Like Peptide 1; Cholecystokinin; Magnetic Resonance Imaging
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood to determine hormonal parameters (gut hormones and reproductive hormones) and the presence of the gene TaqIA1.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lean women: BMI 18-25, weight in kg / height in m2
- Obese women: BMI 30-35, weight in kg / height in m2

SUMMARY:
The purpose of this study is to better understand how female sex hormones influence the food intake in the gut system through the release of satiety hormones as well as through central regulative mechanisms in the brain that subsequently contribute to the control of eating in healthy women at different stages of the ovarian cycle.

DETAILED DESCRIPTION:
Obesity and the associated severe consequences for health, i.e. cardiovascular diseases or Diabetes Type 2 reach the world-wide level of an epidemic with excessive eating as major cause of this development. Study results of veterinary physiology as well as in women let assume that steroid hormones, such as estrogen or progesterone are highly involved in the regulation of eating behavior and the female body weight. This connection is underpinned with the fact that prevalence of adiposity is increased in women in comparison to men in the United States, Switzerland and further countries. A better understanding of the underlying regulatory mechanisms, which in turn influence the food intake in the gut system through the release of satiety hormones as well as through central regulative mechanisms in the brain, provides important foundation in long-term development of new prophylactic and therapeutic options in reduction and prevention of obesity. This gets even more important, as current therapeutic options - beside bariatric surgery - could only show limited success.

Satiety is a process in the brain that leads to a meal being ended, whereby the ingested food causes a reflexive negative feedback mechanism. This mechanism is both fundamentally and specifically in the acute situation strongly influenced through subjective parameters, e.g. eating desires, socio-cultural factors, current social circumstances and individual relation towards eating. Furthermore, food intake is also influenced by genetic factors, whereas e.g. TaqIA1 allele is known to be associated with obesity. According to current knowledge, regulation takes place on peripheral as well as on central level, whereas not only steroid hormones but also satiety hormones - especially cholecystokinin (CCK) and glucagon-like peptide-1 (GLP-1) - are involved on both levels.

The current study aims to examine the connection of steroid hormones, gastrointestinal satiety hormones and neuronal activity in the brain through fMRI. Through the obtained data, the interaction between defined hormone constellations, gastrointestinal satiety hormones and the activation of specific brain areas in obese and normal-weight women should be evaluated. The study design involves the comparison of subjective, hedonic evaluation of different flavoured liquids with different caloric content each through a rating scale as well as objective peripheral (release of CCK and GLP-1) and central (activation of involved brain centres through fMRI) regulation processes in fasted and fed condition of each woman in the two study groups (obese and normal-weighted) in late follicular compared with the luteal phase of ovarian cycle.

ELIGIBILITY:
Inclusion Criteria:

* Physically and psychiatrically healthy women
* Stable body weight (no changes ≥ 5 kg in past year)
* Age 18-35 years
* Regular menses (26-32 d cycles)
* Right-handed
* German language fluency
* Signed informed consent

Exclusion Criteria:

* Life history of eating disorders
* Aversion to the test foods
* Pacemaker or neurostimulator
* Hearing aid
* Surgery to head or heart
* Potential metal parts in body (pacemakers, metal splinters, gun wounds, shrapnel or surgical clips)
* Neurological or psychiatric problems or serious brain injury (such as alcohol or drug abuse, depression, schizophrenia, bipolar disorders, anxiety disorder, claustrophobia, Parkinson's disease, multiple sclerosis, epilepsy)
* High blood pressure, low blood pressure, history of heart disease, irregular heart rate
* Emphysema, chest or respiratory problems (including difficulty breathing through the nose)
* Pregnancy, nursing or pregnancy planned in next three months
* History of gall bladder disease or symptoms (right upper abdominal quadrant pain after meals)
* Polycystic ovary syndrome, as gauged by testosterone levels
* Allergy or sensitivity to lactose
* Allergy to quinine
* Current or previous malignancies
* History of difficult blood sampling

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal-weight and obese women with regular menstrual cycles.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
fMRI responses to food cues | 90 min per study day
  Change in blood oxygen dependent signal (BOLD) in exposure to visual food cues will be measured during a fMRI scan and the difference between responses in the fed condition compared with those in the fasted condition
Change in CCK (satiety hormone) response curve | 30 min per study day
  Blood samples will be collected at 0, 5, 10, 15, 20, 25, 30 min following the ingestion of the meal at each experimental visit, giving a specific curve and analyzed to determine the gut hormone responses. The results will be compared between fast and fed condition, between obese and normal weight women and depending on ovarian cycle phase.
Change in GLP-1 (satiety hormone) response curve | 30 min per study day
  Blood samples will be collected at 0, 5, 10, 15, 20, 25, 30 min following the ingestion of the meal at each experimental visit, giving a specific curve and analyzed to determine the gut hormone responses. The results will be compared between fast and fed condition, between obese and normal weight women and depending on ovarian cycle phase.

SECONDARY OUTCOMES:
Change in food preference indicating motivation to purchase food items | 20 min per study day
  The willingness-to-pay task measures the motivation to obtain food on a gLMS scale. The results will be compared between fast and fed condition, between obese and normal weight women and depending on ovarian cycle phase.
Change in food preference indicating motivation to exert effort | 20 min per study day
  The willingness-to-exert-effort task measures the motivation to obtain food on a gLMS scale. The results will be compared between fast and fed condition, between obese and normal weight women and depending on ovarian cycle phase.
Dietary intake | 30 min per study day
  Measure of the calorie intake
Hedonic ratings | 20 min per study day
  Subjective ratings of flavor pleasantness will be collected using psychophysical rating scales (gLMS)
Subjective sensory ratings | 20 min per study day
  Subjective ratings of hunger sensation will be collected using psychophysical rating scales (gLMS)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Leeners, MD, Principal Investigator — Clinic for Reproductive Endocrinology, University Hospital Zurich; Loredana Asarian, Phd, Study Chair — Institute of Veterinary Physiology, Universirty of Zurich; Philippe Tobler, Prof, Study Chair — Department of Economics, University of Zurich
Locations (1):
- Clinic for Reproductive Endocrinology, University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No